CLINICAL TRIAL: NCT06697509
Title: Improved Detection of Myocardial Fibrosis: a CMR Study
Brief Title: Improved Detection of Myocardial Fibrosis: a Cardiovascular Magnetic Resonance Imaging Study
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Siri Lagethon Heck, Associate professor and consultant radiologist, University Hospital, Akershus
Other Study IDs: 452039
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Myocardial Diseases
Keywords: CMR; Myocardial fibrosis; Biomarkers; Cardiovascular Magnetic Resonance Imaging
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be obtained by venipuncture by dedicated study personnel in relation to the routine pre-procedural clinical examination conducted the same day or the day before the cardiovascular magnetic resonance (CMR) examination
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with suspected or established myocardial disease referred for CMR: Consenting adult patients with suspected or established myocardial disease referred for cardiovascular magnetic resonance (CMR) imaging with gadolinium contrast at Akershus University Hospital

SUMMARY:
Myocardial fibrosis, or scarring, is a common endpoint in many cardiomyopathies and is associated with adverse outcomes, and precise tools to measure myocardial fibrosis are needed. Focal and diffuse myocardial fibrosis can be diagnosed by cardiovascular magnetic resonance (CMR) imaging. However, the CMR procedure is complex and time-consuming and require the use of intravenous gadolinium based contrast agents. A wide range of biomarkers have been associated with the diagnosis and prognosis of cardiovascular disease. In the current study the investigators will assess whether novel and established circulating myocardial biomarkers associate with myocardial fibrosis assessed by CMR. The investigators will also assess whether novel or improved CMR sequences as well as machine learning algorithms improve image quality and the detection of myocardial fibrosis.

DETAILED DESCRIPTION:
This is an observational study of adult patients with suspected myocardial disease referred to cardiovascular magnetic resonance (CMR) with gadolinium contrast. The goal of the study is to assess whether novel and established circulating myocardial biomarkers associate with myocardial fibrosis assessed by CMR. The investigators will also assess novel techniques for detecting myocardial fibrosis by CMR. The plan is to include 1000 patients prior to CMR at Akershus University Hospital.

Blood samples for biomarker measurement will be obtained at the time of CMR. Image quality of novel CMR sequences will be recorded. The diagnostic results of the CMR will be compared to the levels of selected circulating biomarkers of myocardial injury and fibrosis. Novel sequences and techniques for assessing myocardial fibrosis by CMR will be compare to established techniques. Patients will be followed for a minimum of 12 months and the incidence of cardiovascular death, all-cause mortality, acute coronary syndromes, revascularization, heart failure, stroke and cardiac arrhythmias requiring rehospitalization will be recorded. Long-term follow-up information will be obtained from relevant registries

ELIGIBILITY:
Inclusion Criteria:

Consecutive adult patients referred for clinically indicated cardiovascular magnetic resonance (CMR) imaging with gadolinium contrast at Akershus University Hospital will be invited to participate.

Exclusion Criteria:

Participants with contraindication for gadolinium contrast or inability to consent will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational study of patients with suspected myocardial disease referred to in-patient or out-patient cardiovascular magnetic resonance (CMR) examination with gadolinium contrast
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
The presence of focal or diffuse myocardial fibrosis | Baseline
  Focal myocardial fibrosis assessed by late gadolinium enhancement (LGE) and diffuse myocardial fibrosis assessed by the extracellular volume fraction (ECV) by cardiovascular magnetic resonance (CMR) imaging

SECONDARY OUTCOMES:
Composite of cardiovascular death and major adverse cardiac events (MACE) | Up to seven years
  Prognostic endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Akershus University Hospital, Lørenskog, Norge, Norway

IPD SHARING:
Plan to Share IPD: No
Data from the study cannot be publicly shared because of the risk for violating privacy, as regulated by the institutional data protection officer.